CLINICAL TRIAL: NCT03389867
Title: An Open Label Study to Evaluate the Effect of Kaempferia Parviflora in Support of Erectile Function and Male Sexual Health Among Overall Healthy Males 50-70.
Brief Title: Open Label Study to Evaluate the Effect of Kaempferia Parviflora in Support of Erectile Function and Male Sexual Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CL073
Record Dates: First submitted 2017-12-05; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Erectile Function
Keywords: Male sexual health; Erectile function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Male Sexual Health Formulation (Experimental): Kaempferia parviflora extract 100mg daily
  Interventions: Dietary Supplement: Kaempferia parviflora extract

INTERVENTIONS:
Dietary Supplement: Kaempferia parviflora extract
  Other Names: KaempMax™

SUMMARY:
The purpose of this study was to evaluate the overall efficacy and safety of Kaempferia parviflora in overall healthy male human subjects.

DETAILED DESCRIPTION:
This study was an open label safety and efficacy study. Each subject received a specific dose of a formulation containing Kaempferia parviflora. There would be attempted telephone or e-mail contact in 2 weeks following enrollment.

Participants would undergo assessments of blood tests, vital signs, body weight with completion of questionnaires.

The primary objective was to assess the effect of Kaempferia parviflora on erectile function among overall healthy males age 50 to 70.

ELIGIBILITY:
Primary Inclusion Criteria:

1. Healthy male volunteers between the age of 50-70 inclusive
2. Having been (or attempted to be) sexually active for at least the last 6 months
3. Having been in a stable sexual relationship for the past 6 months or more
4. Be able to comply with a 14-day washout period of all sexual performance enhancing medications, nutritional supplements or herbs prior to Day 1 randomization
5. Be able to comply with a 14-day washout period of all nutritional supplements that may contain any of the components of the formulation prior to Day 1 enrollment

Primary Exclusion Criteria:

1. Having a Body Mass Index greater than 34.9
2. Currently receiving or having received treatment in the past 6 months for any sexual disorder or dysfunction (including treatment for erectile function, intercourse satisfaction, orgasmic function, or sexual desire)
3. Attain a score of < 16 on the IIEF-5 questionnaire
4. Primary diagnosis of another sexual disorder (e.g., premature ejaculation)
5. Currently taking supplements including Kaempferia parviflora, DHEA (Dehydroepiandrosterone), chrysin, pregnenolone, grape seed extract, bitter orange, country mallow, ephedra, bitter melon, catuaba, horny goat weed, mucuna pruriens, maca, tribulus terrestris, muira puama, yohimbe or sativa, fenugreek, tongkat ali, Activali, Eurycoma longifolia Jack and goat's rue or any other supplement which has effects on sexual health. Also, testosterone and aromatase inhibitors (letrozole, anastrozole, exemestane, tesolactone) and phosphodiesterase type 5 inhibitors (e.g. sildenafil, tadalafil, vardenafil) unless willing to washout 14 days prior to baseline
6. Having any of the following disorders: benign prostatic hyperplasia (BPH), diabetes mellitus, cancer (including prostate and male breast cancer), insomnia, sleep apnea, heart disease, hypertension, renal disease, liver disease, vascular disease, endocrine abnormalities (e.g. hypogonadism or hypo/hyperthyroidism), multiple sclerosis, psychiatric disorder, acute genitourinary disorder, history of spinal cord injury, herniated disc, penile injury or disease (e.g. Peyronie's disease, priapism or genital anatomic abnormalities) or any other significant medical or surgical procedure that precludes participation in the judgment of the investigator/sub-investigator
7. Currently taking medications for benign prostatic hyperplasia (e.g. tamsulosin, dutasteride, finasteride, terazosin), theophylline medications, antihypertensive medications (e.g. diuretics, sympatholytics, beta blockers, calcium channel blockers), antidiabetic medications, psychiatric medications (e.g. antipsychotic agents, antidepressants, or anxiolytic agents), androgenic and antiandrogenic medications, digitalis, histamine H2-receptor blockers, ketoconazole, niacin, MAOI (monoamine oxidase inhibitor) (e.g. phenelzine), phenobarbital, phenytoin, anticoagulants (e.g. warfarin, high dose aspirin, cilostazol [Pletal], clopidogrel [Plavix], dalteparin [Fragmin], enoxaparin [Lovenox], heparin, ticlopidine [Ticlid]) or receiving nitrate therapy -
8. Laboratory: bilirubin > 2 x ULN (Upper limit of normal) , AST/SGOT (aspartate aminotransferase/serum glutamic oxaloacetic transaminase) and ALT/SGPT (alanine aminotransferase/serum glutamic pyruvic transaminase) ( > 2 x ULN, serum creatinine > 1.5 mg/dL, total cholesterol > 347.9mg/dl, triglycerides > 300mg/dl, and PSA > 4 ng/mL

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 14 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2015-11-29 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
IIEF (International Index of Erectile Dysfunction) questionnaire scores | 30 days
  Mean change in IIEF scores. There are five specific areas addressed including Erectile Function (questions:1-5 & 15;score range: 0-5, maximum score:30); Orgasmic Function (questions:9-10; score range:0-5; maximum score:10); Sexual desire (questions:11-12; score range:1-5; maximum score:10); Intercourse satisfaction (questions:6-8; score range:0-5; maximum score:15); Overall satisfaction (questions:13-14; score range:1-5; maximum score:10). The lower the score represents greater dysfunction within each domain.

SECONDARY OUTCOMES:
GAQ (Global Assessment Question) | 30 days
  Response (yes or no) from Global Assessment Question
Levels of Free Testosterone | 30 days
  Mean change in Free Testosterone levels in pg/ml
Levels of Total Testosterone | 30 days
  Mean change in Total Testosterone levels in ng/dl
Levels of Estradiol | 30 days
  Mean change in Estradiol levels in pg/ml
Levels of DHEA-S | 30 days
  Mean change in DHEA-S levels in ug/dl
Levels of PSA | 30 days
  Mean change in PSA levels in ng/ml
Levels of Total Cholesterol | 30 days
  Mean change in Total Cholesterol levels in mg/dl
Levels of LDL Cholesterol | 30 days
  Mean change in LDL Cholesterol levels in mg/dl
Levels of HDL Cholesterol | 30 days
  Mean change in HDL Cholesterol levels in mg/dl
Levels of Triglycerides | 30 days
  Mean change in Triglyceride levels in mg/dl
Body Mass Index | 30 days
  Mean change in body mass index in kg/m^2 calculated by formula using the body weight (lb.) and the height (in.)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joyal, Principal Investigator — Life Extension

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayta IA, McKinlay JB, Krane RJ. The likely worldwide increase in erectile dysfunction between 1995 and 2025 and some possible policy consequences. BJU Int. 1999 Jul;84(1):50-6. doi: 10.1046/j.1464-410x.1999.00142.x. PMID 10444124
- [Background] Chivapat S, Chavalittumrong P, Attawish A et al. Chronic Toxicity Study of Kaempferia parviflora Wall ex. Extract. Thai J Vet. Med. 40(4):377-383, 2010.
- [Background] . Report from Tokiwa Phytochemical Co. LTD. Sirtmax® PCT/JP2012/084000.
- [Background] Shabsigh R, Anastasiadis AG. Erectile dysfunction. Annu Rev Med. 2003;54:153-68. doi: 10.1146/annurev.med.54.101601.152212. Epub 2002 Aug 19. PMID 12525671
- [Background] Sudwan P, Saenphet K, Saenphet S, Suwansirikul S. Effect of Kaempferia parviflora Wall. ex. Baker on sexual activity of male rats and its toxicity. Southeast Asian J Trop Med Public Health. 2006;37 Suppl 3:210-5. PMID 17547083
- [Background] Sutthanut K, Sripanidkulchai B, Yenjai C, Jay M. Simultaneous identification and quantitation of 11 flavonoid constituents in Kaempferia parviflora by gas chromatography. J Chromatogr A. 2007 Mar 2;1143(1-2):227-33. doi: 10.1016/j.chroma.2007.01.033. Epub 2007 Jan 13. PMID 17266972
- [Background] Tambi MI, Imran MK, Henkel RR. Standardised water-soluble extract of Eurycoma longifolia, Tongkat ali, as testosterone booster for managing men with late-onset hypogonadism? Andrologia. 2012 May;44 Suppl 1:226-30. doi: 10.1111/j.1439-0272.2011.01168.x. Epub 2011 Jun 15. PMID 21671978
- [Background] Tep-Areenan P, Sawasdee P, Randall M. Possible mechanisms of vasorelaxation for 5,7-dimethoxyflavone from Kaempferia parviflora in the rat aorta. Phytother Res. 2010 Oct;24(10):1520-5. doi: 10.1002/ptr.3164. PMID 20878704
- [Background] Wannanon P, Wattanathorn J, Tong-Un T et al. Efficacy Asssessment of Kaempferia Parviflora for the Management of Erectile Dysfunction. OnLine Journal of Biological Sciences. 12 (4), 149-155, 2012
- [Background] Wattanapitayakul SK, Suwatronnakorn M, Chularojmontri L, Herunsalee A, Niumsakul S, Charuchongkolwongse S, Chansuvanich N. Kaempferia parviflora ethanolic extract promoted nitric oxide production in human umbilical vein endothelial cells. J Ethnopharmacol. 2007 Apr 4;110(3):559-62. doi: 10.1016/j.jep.2006.09.037. Epub 2006 Oct 13. PMID 17113256
- [Background] Wattanathorn J, Muchimapura S, Tong-Un T, Saenghong N, Thukhum-Mee W, Sripanidkulchai B. Positive Modulation Effect of 8-Week Consumption of Kaempferia parviflora on Health-Related Physical Fitness and Oxidative Status in Healthy Elderly Volunteers. Evid Based Complement Alternat Med. 2012;2012:732816. doi: 10.1155/2012/732816. Epub 2012 Jul 31. PMID 22899957
- [Background] Wattanathorn J, Pangphukiew P, Muchimapura S et al Aphrodisiac Activity of Kaempferia parviflora. American Journal of Agricultural and Biological Sciences. 7(2);114-120, 2012
- [Derived] Stein RA, Schmid K, Bolivar J, Swick AG, Joyal SV, Hirsh SP. Kaempferia parviflora ethanol extract improves self-assessed sexual health in men: a pilot study. J Integr Med. 2018 Jul;16(4):249-254. doi: 10.1016/j.joim.2018.05.005. Epub 2018 May 26. PMID 29880257
- See also: Kaempferia parviflora — http://www.wantitall.co.za/Health-and-Personal-Care/Kaempferia-Parviflora-60-capsules__B006JXOOT0